CLINICAL TRIAL: NCT06265311
Title: Practical Value of IDUS in Patients With High Risk of Recurrence of Common Bile Duct Stones After ERCP Lithotomy
Brief Title: IDUS in CBD Stone Recurrence High Risk Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zhao Hang, Director of Department of Gastroenterology, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20221307-2
Record Dates: First submitted 2022-12-06; First posted 2024-02-20 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-02

CONDITIONS: Choledocholithiasis; Cholangiopancreatography, Endoscopic Retrograde; Ultrasonography
Keywords: Choledocholithiasis; Cholangiopancreatography, Endoscopic Retrograde; Ultrasonography; Bile Ducts
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDUS examination during ERCP (Experimental): CBD stones cases with high recurrence risks apply IDUS during ERCP
  Interventions: Procedure: IDUS examination
- Control (No Intervention): CBD stones cases with high recurrence risks don't apply IDUS during ERCP

INTERVENTIONS:
Procedure: IDUS examination — for patients with high risks of bile duct stones recurrence using IDUS during ERCP
  Arms: IDUS examination during ERCP

SUMMARY:
This study is designed to observed CBD stones cases with high recurrence risks applying IDUS or not during ERCP.

Patients with CBD stone high recurrence risks were enrolled in this study, and prospectively randomized into IUDS group and control group during lithotomy.

Operation time, radiation time, hospitalization cost, retain of nasobiliary tube, deployment of stent were recorded.

Symptoms and conditions after ERCP were also followed up including blood amylase, routine blood test, abdominal pain, post-ERCP pancreatitis, resection of gallbladder, recurrence of CBD stone and onset of cholangitis.

DETAILED DESCRIPTION:
Patients with CBD stone high recurrence risks were enrolled in this study, and prospectively randomized into IUDS group and control group during lithotomy.

High risks were defined as diameter of CBD>1.5cm, number of calculi>2, and lithotripsy.

Operation time, radiation time, hospitalization cost, retain of nasobiliary tube, deployment of stent were recorded.

Symptoms and conditions after ERCP were also followed up including blood amylase, routine blood test, abdominal pain, post-ERCP pancreatitis, resection of gallbladder, recurrence of CBD stone and onset of cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* 1.Clinical diagnosis of common bile duct stones 2.At least one of the following, diameter of CBD>1.5cm, or number of calculi>2, or lithotripsy during ercp

Exclusion Criteria:

* 1. Clinical diagnosis of liver or biliary malignant tumor. 2. Clinical diagnosis of duodenal malignant tumor 3. Failure or unexpected termination of ERCP 4. Surgery history of gallbladder or bile duct.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
recurrence of bile duct stone or cholangitis | 48 weeks
  patients will be followed up for 48 weeks to record the recurrence of CBD stones or cholangitis
need for a nasobiliary tube | 2 weeks
  it's a Yes or No categorical variable to describe if the patient was placed a nasobiliary tube during ERCP
need for stents | 4 weeks
  it's a Yes or No categorical variable to describe if stents were deployed during ERCP

SECONDARY OUTCOMES:
operation time | intraoperative
  the time from tracheal intubation to the end of ERCP was recorded
radiation time | 4 weeks
  radiation time of each patient was recorded
hospitalization cost | 8 weeks
  hospitalization cost of each patient was recorded
Questionnaire of Symptoms and conditions after ERCP | 8 weeks
  Questionnaire of symptoms and conditions after ERCP were recorded. Degree of abdominal pain and distension were recorded with a highest level of three points respectively.
White blood cell count | 12 weeks
  Routine blood test
Red blood cell count | 12 weeks
  Routine blood test
Platelet count | 12 weeks
  Routine blood test
total bilirubin, direct bilirubin | 12 weeks
  Liver function test
Liver function test (ALT, AST) | 12 weeks
albumin | 12 weeks
  Liver function test
total protein | 12 weeks
  Liver function test
Gamma-glutamyl transferase (GGT) test | 12 weeks
  Liver function test
An alkaline phosphatase (ALP) test | 12 weeks
  Liver function
whether have a resection of gallbladder checklist | 48 weeks
  whether the patient has a resection of gallbladder after ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Hang Zhao, PhD, Principal Investigator — Shanghai Municipal Traditional Chinese Medicine Hospital
Locations (1):
- Shang General Hospital, Shanghai, China